CLINICAL TRIAL: NCT01261325
Title: A Randomized, Double-blind, Placebo-controlled, Multicenter, Parallel-group Study to Evaluate the Efficacy and Safety of Brivaracetam in Subjects (≥16 to 80 Years Old) With Partial Onset Seizures
Brief Title: Brivaracetam Efficacy and Safety Study in Subjects With Partial Onset Seizures
Acronym: BRITE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: N01358; 2010-019361-28 (EudraCT Number)
Expanded Access: NCT03532516 (Available)
Record Dates: First submitted 2010-12-09; First posted 2010-12-16 (Estimated); Results first posted 2016-08-15 (Estimated); Last update posted 2022-07-22 (Actual); Status verified 2022-07

CONDITIONS: Epilepsy
Keywords: Epilepsy; Brivaracetam; Partial Onset Seizures; Adjunctive treatment
MeSH Terms: conditions — Epilepsy | interventions — brivaracetam; Anticonvulsants

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): Matching placebo tablets administered twice daily
  Interventions: Drug: Placebo; Drug: Antiepileptic drugs with market authorization available per country
- Brivaracetam 100 mg/ day (Experimental): Brivaracetam 50 mg/ day administered twice daily.
  Interventions: Drug: Brivaracetam; Drug: Antiepileptic drugs with market authorization available per country
- Brivaracetam 200 mg/ day (Experimental): Brivaracetam 100 mg/ day administered twice daily
  Interventions: Drug: Brivaracetam; Drug: Antiepileptic drugs with market authorization available per country

INTERVENTIONS:
Drug: Placebo — Daily oral dose of two equal intakes of placebo in a double-blinded way for the 12-week treatment period
  Arms: Placebo
Drug: Brivaracetam — Daily oral dose of two equal intakes of Brivaracetam 100 mg/ day in a double-blinded way for the 12-week treatment period
  Arms: Brivaracetam 100 mg/ day
Drug: Brivaracetam — Daily oral dose of two equal intakes of Brivaracetam 200 mg/ day in a double-blinded way for the 12-week treatment period.
  Arms: Brivaracetam 200 mg/ day
Drug: Antiepileptic drugs with market authorization available per country

SUMMARY:
This study will evaluate the efficacy and safety of brivaracetam at doses of 100 and 200mg/day compared to placebo as adjunctive treatment in adult focal epilepsy subjects with partial onset seizures not fully controlled despite current treatment with 1 or 2 concomitant antiepileptic drugs.

ELIGIBILITY:
Inclusion Criteria:

* Well-characterized focal epilepsy/epileptic syndrome according to the 1989 International League Against Epilepsy (ILAE) classification
* Presence of an EEG reading compatible with the clinical diagnosis of focal epilepsy within the last 5 years
* Presence of a brain MRI/computed tomography (CT) scan performed within the last 2 years
* Subjects having at least 8 Type I seizures [POS; focal seizures (according to the 1981 ILAE classification)] during the 8-week Baseline Period with at least 2 Type I seizures during each 4-week interval of the Baseline Period
* Subjects having at least 2 partial onset seizures whether or not secondarily generalized per month during the 3 months preceding V1
* Subjects being uncontrolled while treated by 1 or 2 permitted concomitant AED(s). Vagal Nerve Stimulation (VNS) is allowed and will be counted as a concomitant AED
* Permitted concomitant AED(s) and VNS being stable and at optimal dosage for the subject from at least 1 month (3 months for phenobarbital, phenytoin, and primidone) before V1 and expected to be kept stable during the Baseline and Treatment Period. Benzodiazepine taken more than once a week (for any indication) will be considered as a concomitant AED

Exclusion Criteria:

* Subject previously randomized within this study or any other prior study with BRV as a dosing arm
* Seizure type IA (1981 ILAE classification) nonmotor as only seizure type.
* Subject is currently treated with LEV or has taken LEV within 90 days prior to V1
* Subject has any medical or psychiatric condition, obvious cognitive impairment or mental retardation that, in the opinion of the Investigator, could jeopardize or would compromise the subject's ability to participate in this study
* Subjects whose seizures could not be reliably counted on a regular basis due to their fast and repetitive occurrence (clusters or flurries)
* Subject has history or presence of status epilepticus during the year preceding V1 or during Baseline
* Subject has history or presence of known psychogenic nonepileptic seizures
* Subject on felbamate with less than 18 months exposure before V1
* Subject currently on vigabatrin. Subject with history of vigabatrin use but either no visual fields examination report available including standard static (Humphrey or Octopus) or kinetic perimetry (Goldman) or results of these examinations are abnormal
* Subject taking any drug with possible central nervous system (CNS) effects except if stable from at least 1 month before V1 and expected to be kept stable during the Treatment Period
* Subject has history of cerebrovascular accident, including transient ischemic attack, in the last 6 months
* Subject is suffering from severe cardiovascular disease or peripheral vascular disease
* Subject has a lifetime history of suicide attempt or has suicidal ideation in the past 6 months
* Subject has ongoing psychiatric disease other than mild controlled disorder

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 768 (Actual)
Dates: Start 2010-12; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (207):
- United States (61):
  - 001, Phoenix, Arizona
  - 013, Phoenix, Arizona
  - 006, Tucson, Arizona
  - 775, Little Rock, Arkansas
  - 045, Sacramento, California
  - 025, San Francisco, California
  - 060, Aurora, Colorado
  - 085, Colorado Springs, Colorado
  - 071, Miami, Florida
  - 110, Miami, Florida
  - 073, Naples, Florida
  - 090, Ocala, Florida
  - 027, Orlando, Florida
  - 064, Port Charlotte, Florida
  - 044, Sarasota, Florida
  - 023, Atlanta, Georgia
  - 063, Atlanta, Georgia
  - 062, Columbus, Georgia
  - 048, Rome, Georgia
  - 039, Boise, Idaho
  - 005, Peoria, Illinois
  - 017, Winfield, Illinois
  - 020, Ames, Iowa
  - 069, Iowa City, Iowa
  - 780, Lexington, Kentucky
  - 092, Hammond, Louisiana
  - 008, Bethesda, Maryland
  - 068, Waldorf, Maryland
  - 055, East Lansing, Michigan
  - 009, Golden Valley, Minnesota
  - 051, Missoula, Montana
  - 032, Lebanon, New Hampshire
  - 042, Hamilton, New Jersey
  - 058, Voorhees Township, New Jersey
  - 095, Kingston, New York
  - 022, New York, New York
  - 099, New York, New York
  - 098, Poughkeepsie, New York
  - 010, Asheville, North Carolina
  - 003, Durham, North Carolina
  - 096, Canton, Ohio
  - 034, Cleveland, Ohio
  - 070, Columbus, Ohio
  - 002, Toledo, Ohio
  - 043, Oklahoma City, Oklahoma
  - 091, Oklahoma City, Oklahoma
  - 054, Tulsa, Oklahoma
  - 015, Philadelphia, Pennsylvania
  - 028, Charleston, South Carolina
  - 021, Port Royal, South Carolina
  - 050, Arlington, Texas
  - 061, Austin, Texas
  - 011, Dallas, Texas
  - 035, Dallas, Texas
  - 049, Houston, Texas
  - 036, Charlottesville, Virginia
  - 033, Seattle, Washington
  - 056, Spokane, Washington
  - 052, Madison, Wisconsin
  - 057, Milwaukee, Wisconsin
  - 089, Casper, Wyoming
- Austria (4):
  - 202, Innsbruck
  - 201, Linz
  - 200, Vienna
  - 203, Vienna
- Belgium (3):
  - 226, Hechteleksel
  - 227, Leuven
  - 228, Liège
- Brazil (4):
  - 104, Belo Horizonte
  - 100, Florianópolis
  - 103, Riberao Preto
  - 101, São Paulo
- Bulgaria (3):
  - 294, Blagoevrad
  - 286, Sofia
  - 287, Sofia
- Canada (6):
  - 075, Calgary, Alberta
  - 078, London, Ontario
  - 076, Toronto, Ontario
  - 077, Greenfield Park, Quebec
  - 079, Montreal, Quebec
  - 080, Saskatoon, Saskatchewan
- Czechia (7):
  - 916, Kroměříž
  - 251, Ostrava
  - 256, Ostrava
  - 913, Ostrava Poruba
  - 252, Prague
  - 253, Prague
  - 250, Zlín
- Estonia (4):
  - 650, Tallinn
  - 652, Tallinn
  - 653, Tallinn
  - 651, Tartu
- Finland (4):
  - 275, Kuopio
  - 278, Oulu
  - 276, Tampere
  - 277, Turku
- France (3):
  - 301, Béthune
  - 308, Marseille
  - 305, Montpellier
- Germany (12):
  - 329, Berlin
  - 326, Bernau
  - 332, Bielefeld
  - 902, Erlangen
  - 331, Göttingen
  - 904, Kehl-Kork
  - 327, Kiel
  - 900, Marburg
  - 335, München
  - 334, Osnabrück
  - 330, Ravensburg
  - 328, Ulm
- Hong Kong (2):
  - 701, Hong Kong
  - 700, Shatin
- Hungary (5):
  - 410, Budapest
  - 411, Budapest
  - 412, Budapest
  - 414, Debrecen
  - 413, Kecskemét
- India (6):
  - 727, Hyderabad, Andhra Pradesh
  - 725, Mumbai, Maharashtra
  - 728, Mumbai, Maharashtra
  - 731, Nashik, Maharashtra
  - 726, Bangalore
  - 729, Madurai
- Italy (10):
  - 377, Monserrato, Cagliari
  - 378, Bari
  - 380, Florence
  - 379, Milan
  - 386, Napoli
  - 376, Perugia
  - 375, Pisa
  - 383, Pozzilli
  - 384, Reggio Calabria
  - 382, Torino
- Japan (5):
  - 855, Hiroshima
  - 852, Itami
  - 850, Osaka
  - 851, Shizuoka
  - 854, Yokohama
- Latvia (5):
  - 627, Daugapils
  - 629, Jēkabpils
  - 626, Riga
  - 628, Riga
  - 625, Valmiera
- Lithuania (3):
  - 425, Alytus
  - 427, Kaunas
  - 426, Vilnius
- Mexico (6):
  - 126, Guadalajara, Jalisco
  - 128, Guadalajara, Jalisco
  - 129, Aguascalientes
  - 127, Culiacán
  - 125, Distrito Federal
  - 130, Mexico City
- Netherlands (3):
  - 401, Heemstede
  - 400, Heeze
  - 403, Zwolle
- Poland (13):
  - 475, Bialystok
  - 485, Gdansk
  - 791, Gdansk
  - 478, Katowice
  - 480, Katowice
  - 481, Katowice
  - 476, Krakow
  - 793, Krakow
  - 483, Lublin
  - 477, Poznan
  - 479, Poznan
  - 482, Poznan
  - 488, Warsaw
- 038, San Juan, Puerto Rico
- Russia (7):
  - 501, Kazan'
  - 506, Kazan'
  - 502, Moscow
  - 503, Moscow
  - 505, Moscow
  - 509, Nizhny Novgorod
  - 508, Smolensk
- South Korea (5):
  - 753, Busan
  - 752, Gwangju
  - 750, Seoul
  - 751, Seoul
  - 754, Seoul
- Spain (10):
  - 536, Badalona
  - 528, Barcelona
  - 529, Barcelona
  - 535, Barcelona
  - 540, Barcelona
  - 539, Donostia / San Sebastian
  - 532, Santiago de Compostela
  - 527, Valencia
  - 537, Valencia
  - 526, Valladolid
- Sweden (3):
  - 551, Gothenburg
  - 552, Linköping
  - 550, Stockholm
- Taiwan (4):
  - 806, Kaohsiung City
  - 801, Taichung
  - 800, Tainan
  - 803, Taoyuan Hsien
- United Kingdom (8):
  - 603, Birmingham
  - 606, Cardiff
  - 601, Cornwall
  - 600, London
  - 605, Middlesbrough
  - 607, Newcastle
  - 608, Salford
  - 602, Swansea

REFERENCES:
- [Result] Toledo M, Whitesides J, Schiemann J, Johnson ME, Eckhardt K, McDonough B, Borghs S, Kwan P. Safety, tolerability, and seizure control during long-term treatment with adjunctive brivaracetam for partial-onset seizures. Epilepsia. 2016 Jul;57(7):1139-51. doi: 10.1111/epi.13416. Epub 2016 Jun 6. PMID 27265725
- [Result] Ben-Menachem E, Mameniskiene R, Quarato PP, Klein P, Gamage J, Schiemann J, Johnson ME, Whitesides J, McDonough B, Eckhardt K. Efficacy and safety of brivaracetam for partial-onset seizures in 3 pooled clinical studies. Neurology. 2016 Jul 19;87(3):314-23. doi: 10.1212/WNL.0000000000002864. Epub 2016 Jun 22. PMID 27335114
- [Result] Klein P, Schiemann J, Sperling MR, Whitesides J, Liang W, Stalvey T, Brandt C, Kwan P. A randomized, double-blind, placebo-controlled, multicenter, parallel-group study to evaluate the efficacy and safety of adjunctive brivaracetam in adult patients with uncontrolled partial-onset seizures. Epilepsia. 2015 Dec;56(12):1890-8. doi: 10.1111/epi.13212. Epub 2015 Oct 16. PMID 26471380
- [Result] Brodie MJ, Whitesides J, Schiemann J, D'Souza J, Johnson ME. Tolerability, safety, and efficacy of adjunctive brivaracetam for focal seizures in older patients: A pooled analysis from three phase III studies. Epilepsy Res. 2016 Nov;127:114-118. doi: 10.1016/j.eplepsyres.2016.08.018. Epub 2016 Aug 18. PMID 27589414
- [Result] Moseley BD, Sperling MR, Asadi-Pooya AA, Diaz A, Elmouft S, Schiemann J, Whitesides J. Efficacy, safety, and tolerability of adjunctive brivaracetam for secondarily generalized tonic-clonic seizures: Pooled results from three Phase III studies. Epilepsy Res. 2016 Nov;127:179-185. doi: 10.1016/j.eplepsyres.2016.09.003. Epub 2016 Sep 3. PMID 27608437
- [Result] Brandt C, Borghs S, Elmoufti S, Mueller K, Townsend R, de la Loge C. Health-related quality of life in double-blind Phase III studies of brivaracetam as adjunctive therapy of focal seizures: A pooled, post-hoc analysis. Epilepsy Behav. 2017 Apr;69:80-85. doi: 10.1016/j.yebeh.2016.11.031. Epub 2017 Feb 23. PMID 28236727
- [Result] Klein P, Johnson ME, Schiemann J, Whitesides J. Time to onset of sustained >/=50% responder status in patients with focal (partial-onset) seizures in three phase III studies of adjunctive brivaracetam treatment. Epilepsia. 2017 Feb;58(2):e21-e25. doi: 10.1111/epi.13631. Epub 2016 Dec 18. PMID 27988967
- [Result] Asadi-Pooya AA, Sperling MR, Chung S, Klein P, Diaz A, Elmoufti S, Schiemann J, Whitesides J. Efficacy and tolerability of adjunctive brivaracetam in patients with prior antiepileptic drug exposure: A post-hoc study. Epilepsy Res. 2017 Mar;131:70-75. doi: 10.1016/j.eplepsyres.2017.02.007. Epub 2017 Feb 27. PMID 28279891
- [Result] Benbadis S, Klein P, Schiemann J, Diaz A, Elmoufti S, Whitesides J. Efficacy, safety, and tolerability of brivaracetam with concomitant lamotrigine or concomitant topiramate in pooled Phase III randomized, double-blind trials: A post-hoc analysis. Epilepsy Behav. 2018 Mar;80:129-134. doi: 10.1016/j.yebeh.2017.12.024. Epub 2018 Feb 3. PMID 29414542
- [Result] Brodie MJ, Fakhoury T, McDonough B, Colson AO, Stockis A, Elmoufti S, Whitesides J. Brivaracetam-induced elevation of carbamazepine epoxide levels: A post-hoc analysis from the clinical development program. Epilepsy Res. 2018 Sep;145:55-62. doi: 10.1016/j.eplepsyres.2018.06.002. Epub 2018 Jun 4. PMID 29908435
- [Result] Klein P, Laloyaux C, Elmoufti S, Gasalla T, Martin MS. Time course of 75%-100% efficacy response of adjunctive brivaracetam. Acta Neurol Scand. 2020 Aug;142(2):175-180. doi: 10.1111/ane.13287. Epub 2020 Jun 9. PMID 32432339
- [Result] Moseley BD, Dimova S, Elmoufti S, Laloyaux C, Asadi-Pooya AA. Long-term efficacy and tolerability of adjunctive brivaracetam in adults with focal to bilateral tonic-clonic (secondary generalized) seizures: Post hoc pooled analysis. Epilepsy Res. 2021 Oct;176:106694. doi: 10.1016/j.eplepsyres.2021.106694. Epub 2021 Jun 24. PMID 34218211
- [Result] Ryvlin P, Dimova S, Elmoufti S, Floricel F, Laloyaux C, Nondonfaz X, Biton V. Tolerability and efficacy of adjunctive brivaracetam in adults with focal seizures by concomitant antiseizure medication use: Pooled results from three phase 3 trials. Epilepsia. 2022 Aug;63(8):2024-2036. doi: 10.1111/epi.17304. Epub 2022 Jun 10. PMID 35582748
- [Derived] Brandt C, Dimova S, Elmoufti S, Laloyaux C, Nondonfaz X, Klein P. Retention, efficacy, tolerability, and quality of life during long-term adjunctive brivaracetam treatment by number of lifetime antiseizure medications: A post hoc analysis of phase 3 trials in adults with focal seizures. Epilepsy Behav. 2023 Jan;138:108967. doi: 10.1016/j.yebeh.2022.108967. Epub 2022 Nov 23. PMID 36435010
- [Derived] Bresnahan R, Panebianco M, Marson AG. Brivaracetam add-on therapy for drug-resistant epilepsy. Cochrane Database Syst Rev. 2022 Mar 14;3(3):CD011501. doi: 10.1002/14651858.CD011501.pub3. PMID 35285519
- [Derived] Lee SK, Heo K, Kim SE, Lee SA, Elmoufti S, Laloyaux C, Hur B. Effect of Number of Previous Antiseizure Medications on Efficacy and Tolerability of Adjunctive Brivaracetam for Uncontrolled Focal Seizures: Post Hoc Analysis. Adv Ther. 2021 Jul;38(7):4082-4099. doi: 10.1007/s12325-021-01816-5. Epub 2021 Jun 21. PMID 34155568
- [Derived] Toledo M, Brandt C, Quarato PP, Schulz AL, Cleveland JM, Wagener G, Klein P. Long-term safety, efficacy, and quality of life during adjunctive brivaracetam treatment in patients with uncontrolled epilepsy: An open-label follow-up trial. Epilepsy Behav. 2021 May;118:107897. doi: 10.1016/j.yebeh.2021.107897. Epub 2021 Mar 27. PMID 33780735
- [Derived] Markham A. Brivaracetam: First Global Approval. Drugs. 2016 Mar;76(4):517-22. doi: 10.1007/s40265-016-0555-6. PMID 26899665
- See also: Product Information — https://www.briviact.com/briviact-PI.pdf?v=1479491757
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment for the N01358 study began in December 2010. The study concluded in May 2014.
Pre-assignment Details: The Participant Flow and Baseline Demographics data is taken from the Randomized Set (RS). The RS consists of all subjects who were randomized.
Groups:
- Brivaracetam 100 mg/Day: Brivaracetam 50 mg administered twice daily
- Brivaracetam 200 mg/Day: Brivaracetam 100 mg administered twice daily
Period: Overall Study
Arm/Group | Placebo | Brivaracetam 100 mg/Day | Brivaracetam 200 mg/Day
Started | 263 | 254 | 251
Completed | 246 | 225 | 225
Not Completed | 17 | 29 | 26
Not completed — Lack of Efficacy | 1 | 1 | 0
Not completed — Withdrawal by Subject | 2 | 2 | 4
Not completed — SAE, non-fatal | 1 | 5 | 1
Not completed — AE, non-serious non-fatal | 9 | 15 | 13
Not completed — SAE, non-fatal+AE, non-serious non-fatal | 0 | 1 | 1
Not completed — Non Compliance | 2 | 0 | 0
Not completed — Patient Randomized by Mistake | 0 | 1 | 0
Not completed — Erroneously Randomized | 1 | 0 | 0
Not completed — Screen Failure | 1 | 0 | 0
Not completed — Randomized in Error | 0 | 0 | 1
Not completed — Protocol Violation | 0 | 3 | 1
Not completed — Lost to Follow-up | 0 | 1 | 3
Not completed — AE, serious fatal | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: Baseline Characteristics consist of the Randomized Set (RS). The RS includes all subjects that were randomized.
Arm/Group | Placebo | Brivaracetam 100 mg/Day | Brivaracetam 200 mg/Day | Total Title
Number analyzed (Participants) | 263 | 254 | 251 | 768
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.8 (12.8) | 39.0 (13.4) | 39.7 (12.8) | 39.5 (13.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 128 | 152 | 117 | 397
  Male | 135 | 102 | 134 | 371
Weight [Median (Standard Deviation); unit: kilograms] | 76.1 (19.9) | 74.1 (16.8) | 75.5 (19.0) | 75.2 (18.6)
Height [Mean (Standard Deviation); unit: centimeters] | 168.4 (10.0) | 166.6 (9.8) | 168.7 (9.9) | 167.9 (9.9)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 26.6 (5.7) | 26.7 (5.6) | 26.4 (6.0) | 26.6 (5.8)
Racial Group [Number; unit: participants]
  American Indian or Alaska Native | 10 | 8 | 11 | 29
  Asian | 32 | 32 | 29 | 93
  Black or African American | 11 | 8 | 7 | 26
  White | 190 | 183 | 183 | 556
  Other | 17 | 21 | 18 | 56
  Missing | 3 | 2 | 3 | 8

OUTCOME MEASURES:

1. Primary Outcome: Percent Reduction Over Placebo for Partial Onset Seizure (Type I) Frequency Over the Treatment Period Standardized to a 28-day Duration
Description: Primary endpoint: United States of America (FDA)
Time Frame: 12 week Treatment Period
Population: Analysis population consists of the Intent-to-Treat (ITT) Population, which is all randomized subjects who received at least 1 dose of study medication and have at least 1 post-Baseline seizure diary.
Measure: Number; unit: Percentage of reduction
Arm/Group | Brivaracetam 100 mg/Day | Brivaracetam 200 mg/Day | Placebo
Number analyzed (Participants) | 252 | 249 | 259
Percentage of reduction | 22.8 | 23.2 | 0
Statistical Analysis 1: Comparison: Brivaracetam 100 mg/Day; Test type: Superiority or Other; p < 0.001, ANCOVA — Type I error rate of 0.05 based on a Hochberg multiple comparison procedure would be considered statistically significant" or similar, as accurate and appropriate; Effects of treatment, country, combination of LEV status and number of previous AEDs, and log-transformed baseline seizure frequency are in the model; Percent reduction over PBO = 22.8, 95% CI 2-sided [13.3 to 31.2]
Statistical Analysis 2: Comparison: Brivaracetam 200 mg/Day; Test type: Superiority or Other; p < 0.001, ANCOVA — Statistically significant with control of Type I error rate based on a Hochberg multiple comparison procedure; [statistical method as in outcome 1, analysis 1]; Percent reduction over PBO = 23.2, 95% CI 2-sided [13.8 to 31.6]

2. Primary Outcome: 50% Responder Rate for Partial Onset Seizure (Type I) Frequency Over the Treatment Period Standardized to a 28-day Duration
Description: Primary Endpoint: European Regulatory Authorities A responder is a participant who experienced a 50% or greater reduction in partial onset seizure (Type I) frequency over the Treatment Period standardized to a 28-day duration.
Time Frame: Baseline to 12 week Treatment Period
Population: as for outcome 1
Measure: Number; unit: Percentage of subjects
Arm/Group | Placebo | Brivaracetam 100 mg/Day | Brivaracetam 200 mg/Day
Number analyzed (Participants) | 259 | 252 | 249
Percentage of subjects
  Responders | 21.6 | 38.9 | 37.8
  Non-Responders | 78.4 | 61.1 | 62.2
Statistical Analysis 1: Comparison: Placebo vs Brivaracetam 100 mg/Day; Test type: Superiority or Other; p < 0.001, Regression, Logistic — Statistically significant with control of Type I error rate based on a Hochberg multiple comparison procedure; [statistical method as in outcome 1, analysis 1]; Odds ratio (BRV versus PBO) = 2.39, 95% CI 2-sided [1.6 to 3.6]
Statistical Analysis 2: Comparison: Placebo vs Brivaracetam 200 mg/Day; Test type: Superiority or Other; p < 0.001, Regression, Logistic — Statistically significant with control of Type I error rate based on a Hochberg multiple comparison procedure; [statistical method as in outcome 1, analysis 1]; Odds ratio (BRV versus PBO) = 2.19, 95% CI 2-sided [1.5 to 3.3]

3. Secondary Outcome: Percent Change in Partial Onset Seizure (Type I) Frequency From the Baseline to the Treatment Period
Time Frame: Baseline to 12 week Treatment Period
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: percentage of change
Arm/Group | Placebo | Brivaracetam 100 mg/Day | Brivaracetam 200 mg/Day
Number analyzed (Participants) | 259 | 252 | 249
percentage of change | 17.6 [-8.3 to 46.0] | 37.2 [0.1 to 69.4] | 35.6 [4.8 to 66.2]
Statistical Analysis 1: Comparison: Placebo vs Brivaracetam 100 mg/Day; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney) — Statistically significant at a nominal 0.050 significance level; Median difference vs placebo = 15.8, 95% CI 2-sided [7.6 to 24.2] — Hodges-Lehmann non-parametric effect estimates and corresponding two-sided 95% confidence intervals are provided above
Statistical Analysis 2: Comparison: Placebo vs Brivaracetam 200 mg/Day; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney) — Statistically significant at a nominal 0.050 significance level; Median difference vs placebo = 18.1, 95% CI 2-sided [10.4 to 26.4] — Hodges-Lehmann non-parametric effect estimates and corresponding two-sided 95% confidence intervals are provided above

4. Secondary Outcome: Categorized Percent Reduction Form Baseline in Seizure Frequency for Partial Onset Seizure (Type I) Over the Treatment Period
Time Frame: Baseline to 12 week Treatment Period
Population: as for outcome 1
Measure: Number; unit: percentage of subjects
Arm/Group | Placebo | Brivaracetam 100 mg/Day | Brivaracetam 200 mg/Day
Number analyzed (Participants) | 259 | 252 | 249
percentage of subjects
  <-25 % | 16.6 | 14.3 | 10.8
  -25 % to <25 % | 40.5 | 28.6 | 29.3
  25 % to <50 % | 21.2 | 18.3 | 22.1
  50 % to <75 % | 13.9 | 19.0 | 18.1
  75 % to <100 % | 6.9 | 13.9 | 13.7
  100 % | 0.8 | 6.0 | 6.0

5. Secondary Outcome: Seizure Freedom Rate (All Seizure Types) During the 12-week Treatment Period
Time Frame: 12 week Treatment Period
Population: as for outcome 1
Measure: Number; unit: percentage of subjects
Arm/Group | Placebo | Brivaracetam 100 mg/Day | Brivaracetam 200 mg/Day
Number analyzed (Participants) | 259 | 252 | 249
percentage of subjects
  Seizure free | 0.8 | 5.2 | 4.0
  No seizures but discontinued | 0.4 | 1.2 | 1.2
  Not seizure free | 98.8 | 93.7 | 94.8

6. Secondary Outcome: All Seizure Frequency (Type I + II + III) During the 12-week Treatment Period
Time Frame: 12 week Treatment Period
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: number of seizures/ 28-day
Arm/Group | Placebo | Brivaracetam 100 mg/Day | Brivaracetam 200 mg/Day
Number analyzed (Participants) | 259 | 252 | 249
number of seizures/ 28-day | 8.7 [4.3 to 23.6] | 6.3 [2.7 to 17.8] | 5.8 [2.3 to 14.2]

7. Secondary Outcome: Time to the First Type I Seizure During the Treatment Period
Time Frame: 12 week Treatment Period
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Placebo | Brivaracetam 100 mg/Day | Brivaracetam 200 mg/Day
Number analyzed (Participants) | 259 | 252 | 249
days | 3 [2 to 3] | 5 [3 to 7] | 6 [4 to 7]
Statistical Analysis 1: Comparison: Placebo vs Brivaracetam 100 mg/Day; Test type: Superiority or Other; p < 0.001, Semi-parametric hazards regression model — Statistically significant at a nominal 0.050 significance level; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.67, 95% CI 2-sided [0.56 to 0.82] — Hazard ratio is Brivaracetam versus Placebo
Statistical Analysis 2: Comparison: Placebo vs Brivaracetam 200 mg/Day; Test type: Superiority or Other; p < 0.001, Semi-parametric hazards regression model — Statistically significant at a nominal 0.050 significance level; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.65, 95% CI 2-sided [0.54 to 0.79] — Hazard ratio is Brivaracetam versus Placebo

8. Secondary Outcome: Time to the Fifth Type I Seizure During the Treatment Period
Time Frame: 12 week Treatment Period
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Placebo | Brivaracetam 100 mg/Day | Brivaracetam 200 mg/Day
Number analyzed (Participants) | 259 | 252 | 249
days | 16 [12 to 19] | 21 [17 to 25] | 23 [20 to 26]
Statistical Analysis 1: Comparison: Placebo vs Brivaracetam 100 mg/Day; Test type: Superiority or Other; p < 0.001, Semi-parametric hazards regression model — Statistically significant at a nominal 0.050 significance level; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.65, 95% CI 2-sided [0.53 to 0.80] — Hazard ratio is Brivaracetam versus Placebo
Statistical Analysis 2: Comparison: Placebo vs Brivaracetam 200 mg/Day; Test type: Superiority or Other; p < 0.001, Semi-parametric hazards regression model — Statistically significant at a nominal 0.050 significance level; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.58, 95% CI 2-sided [0.47 to 0.71] — Hazard ratio is Brivaracetam versus Placebo

9. Secondary Outcome: Time to the Tenth Type I Seizure During the Treatment Period
Time Frame: 12 week Treatment Period
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Placebo | Brivaracetam 100 mg/Day | Brivaracetam 200 mg/Day
Number analyzed (Participants) | 259 | 252 | 249
days | 32 [24 to 36] | 37 [29 to 46] | 43 [36 to 49]
Statistical Analysis 1: Comparison: Placebo vs Brivaracetam 100 mg/Day; Test type: Superiority or Other; p = 0.009, Semi-parametric hazards regression model — Statistically significant at a nominal 0.050 significance level; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.75, 95% CI 2-sided [0.60 to 0.93]
Statistical Analysis 2: Comparison: Placebo vs Brivaracetam 200 mg/Day; Test type: Superiority or Other; p < 0.001, Semi-parametric hazards regression model — Statistically significant at a nominal 0.050 significance level; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.68, 95% CI 2-sided [0.55 to 0.85]

ADVERSE EVENTS:
Time Frame: Treatment-emergent Adverse Events (TEAE) were collected during the study up to week 18
Description: TEAEs are comprised of the Safety Population, which consists of all randomized subjects who receive at least 1 dose of study medication.
  The Non-serious Adverse Events section represents a >= 5% threshold of subjects experiencing Non-serious TEAEs in any treatment group and not the total population.
Arm/Group | Placebo | Brivaracetam 100 mg/Day | Brivaracetam 200 mg/Day
Serious Adverse Events (participants affected / at risk) | 9/261 | 8/253 | 8/250
Other Adverse Events (participants affected / at risk) | 61/261 | 96/253 | 97/250
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Placebo (N=261) | Brivaracetam 100 mg/Day (N=253) | Brivaracetam 200 mg/Day (N=250)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Death (General disorders) | 0 (0) | 0 (0) | 1 (1)
Sudden unexplained death in epilepsy (General disorders) | 0 (0) | 0 (0) | 1 (1)
Localised infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Meningitis viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1/231 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 2 (2)
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Traumatic renal injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Thymoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Grand mal convulsion (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Seizure cluster (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Status epilepticus (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Epilepsy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Postictal state (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Adjustment disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Conversion disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Epileptic psychosis (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Psychotic disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=261) | Brivaracetam 100 mg/Day (N=253) | Brivaracetam 200 mg/Day (N=250)
Fatigue (General disorders) | 10 (10) | 19 (19) | 29 (32)
Urinary tract infection (Infections and infestations) | 8 (8) | 13 (13) | 2 (2)
Somnolence (Nervous system disorders) | 20 (20) | 49 (53) | 42 (43)
Dizziness (Nervous system disorders) | 13 (14) | 26 (27) | 36 (38)
Headache (Nervous system disorders) | 22 (30) | 17 (18) | 20 (21)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
UCB has > 60 but <= 180 days to review results communications prior to public release and may delete information that is confidential and compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that the results shall be published regardless of outcome.